CLINICAL TRIAL: NCT06644755
Title: Phase 1, Open-Label, Multicenter, First-In-Human Trial of Ds-2243a in Participants With Advanced Solid Tumors
Brief Title: First-in-Human Trial of DS-2243a in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DS2243-054
Record Dates: First submitted 2024-10-04; First posted 2024-10-16 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Solid Tumors; Sarcoma
Keywords: synovial sarcoma; ny-eso-1; DS-2243a; Myxoid Round cell Liposarcoma; sarcoma; NSCLC; UC; Bladder Cancer; NY-ESO; HLA-A2; Advanced solid tumors
MeSH Terms: conditions — Sarcoma; Sarcoma, Synovial; Liposarcoma, Myxoid; Urinary Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: This is an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1: Dose Escalation DS-2243a (Experimental): Participants will receive DS-2243a at escalating doses. The recommended dose for expansion (RDE) will be calculated using data collected from this population.
  Interventions: Drug: DS-2243a
- Part 2: Dose Expansion SS/MRCLS (Experimental): Participants with synovial sarcoma or myxoid/round cell liposarcoma will receive DS-2243a at the recommended dose for expansion (RDE)
  Interventions: Drug: DS-2243a
- Part 2: Dose Expansion Sq-NSCLC (Experimental): Participants with squamous cell carcinoma-non-small cell lung cancer will receive DS-2243a at the recommended dose for expansion (RDE)
  Interventions: Drug: DS-2243a
- Part 2: Dose Expansion UC (Experimental): Participants with urothelial carcinoma will receive DS-2243a at the recommended dose for expansion (RDE)
  Interventions: Drug: DS-2243a
- Part 2: Dose Expansion Ad-NSCLC (Experimental): Participants with adenocarcinoma-non-small cell lung cancer will receive DS-2243a at the recommended dose for expansion (RDE)
  Interventions: Drug: DS-2243a

INTERVENTIONS:
Drug: DS-2243a — Escalation Part: DS-2243a will be administered at escalating doses to determine the RDE
  Expansion Part: DS-2243a will be administered at RDE

SUMMARY:
This 2-part study will evaluate safety, tolerability, and clinical efficacy of DS-2243a as a treatment for participants with advanced solid tumors.

DETAILED DESCRIPTION:
This is a global, multicenter, open-label, first-in-human, Phase 1 trial of DS-2243a as a treatment for locally advanced or metastatic synovial sarcoma (SS), myxoid/round cell liposarcoma (MRCLS), squamous cell carcinoma type non-small cell lung cancer (Sq-NSCLC), adenocarcinoma type non-small cell lung cancer (Ad-NSCLC), or urothelial carcinoma (UC) participants with HLA-A2 and/or NY-ESO positive. The trial consists of 2 parts: the Dose Escalation Part (Part 1) and the Dose Expansion Part (Part 2).

ELIGIBILITY:
Key Inclusion Criteria:

1. Sign and date the main ICF.
2. Adults ≥18 years at the time the biosample ICF or main ICF, whichever is signed first.

   Follow local regulatory requirements if the legal age of consent for trial participation is >18 years old.
3. One of the following histologically or cytologically documented cancers:

   Advanced (metastatic or unresectable) SS Advanced (metastatic or unresectable) MRCLS Metastatic or unresectable locally advanced NSCLC (Ad/Sq) Metastatic or unresectable locally advanced UC
4. Relapsed from, refractory to, or intolerant to appropriate therapies [eg, standard of care (SOC) therapy] to provide clinical benefit for their condition as assessed by their physician and/or investigator. [For South Korea only: Relapsed from, refractory to, or intolerant to all available therapies (eg, SOC therapy domestically approved) for their condition.]
5. HLA-A*02:01, 02:02, 02:03, 02:04, 02:05, 02:06, 02:09, 02:10, or 02:11 positive.
6. Has measurable disease based on RECIST v1.1 on computed tomography/magnetic resonance imaging (CT/MRI).
7. Is willing and able to provide adequate pre-treatment or archival tumor tissue sample.
8. Has Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0 or 1 at Screening.
9. Meets the following required baseline local laboratory data within 14 days prior to start of trial intervention administration:

   1. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 × upper limit of normal (ULN) in participants with no liver metastasis, or ≤5 × ULN in participants with liver metastasis
   2. Total bilirubin (TBL) ≤1.5 × ULN (≤3 × ULN for participants with a documented history of Gilbert's syndrome)
   3. Absolute neutrophil count (ANC) ≥1.5 × 10^9/L
   4. Platelet count ≥100 × 10^9/L
   5. Hemoglobin ≥8 g/dL
   6. Creatinine clearance (CrCl) ≥45 mL/min as calculated using the Cockcroft-Gault equation (Section 10.3.1)

   Note: Any blood or blood product transfusion is allowed up to 7 days before the hematology evaluations and any dose of hematologic growth factor is allowed up to 14 days before the hematology evaluations.
10. a) A female participant of childbearing potential (CBP), as defined in Section 10.3.5.1, is eligible to participate if the following conditions are met: Participant is not pregnant as confirmed by highly sensitive pregnancy test (see Section 10.3.5.3). Participant does not breastfeed during the trial intervention period and for at least 120 days after last dose of trial intervention. Participant agrees to adhere to a contraceptive method that is highly effective (Section 10.3.5.2) and agrees not to donate eggs (ova, oocytes) to others or freeze/store eggs during the intervention period and for at least the time needed to eliminate the trial intervention after the last dose. The length of time required to continue contraception after last dose for the trial intervention is 120 days. Preservation of eggs may be considered prior to first dose of trial intervention.

    b) A male participant capable of producing sperm is eligible to participate if he agrees to the following during the Treatment Period and for at least the time needed to eliminate the trial intervention. The length of time required to continue contraception after the last dose of the trial intervention is 120 days.
    * Avoid donating sperm. Note: Preservation of sperm should be considered prior to enrollment/randomization in this trial.
    * Adhere to either of the following contraception methods:

      * True abstinence from penile-vaginal intercourse, when this is in line with the preferred and usual lifestyle of the participant, OR
      * Uses a penile/external condom when having penile-vaginal intercourse with a nonparticipant of childbearing potential (see Section 10.3.5) PLUS partner use of an additional contraceptive method (see Section 10.3.5.2), as a condom may break or leak. Contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. If the contraception requirements in the local label for any of the trial interventions are more stringent than the requirements above, the local label requirements are to be followed.

Note: If the participant is azoospermic (vasectomized or secondary to medical cause, documented from the site personnel's review of the participant's medical records, medical examination, or medical history interview), no contraception is required.

Key Exclusion Criteria:

1. Has received prior therapy targeting NY-ESO-1.
2. Has an inadequate treatment washout period prior to the start of trial intervention, defined as follows:

   1. Radiation therapy: <4 weeks (or <2 weeks if palliative radiation therapy without abdominal/pelvic radiation)
   2. Chemotherapy, antibody-based anticancer therapy, immunotherapy: <4 weeks
   3. Small molecules (eg, tyrosine kinase inhibitors): <2 weeks or 5 half-lives, whichever is longer
3. Has known symptomatic central nervous system (CNS) metastases, leptomeningeal disease, or cord compression. Note: Asymptomatic or adequately treated CNS metastases are not exclusionary provided that, in the opinion of the investigator, the participant is neurologically stable.

   MRI/CT of the brain is required for all participants during Screening Period (see Section 8.3.1).
4. Uncontrolled or clinically significant cardiovascular disease, including the following:

   1. Myocardial infarction within 6 months prior to screening
   2. Uncontrolled angina pectoris within 6 months prior to screening
   3. New York Heart Association (NYHA) Class III or IV congestive heart failure
   4. Left ventricular ejection fraction (LVEF) ≤50% or lower than the institutional lower limit of normal
   5. QT interval corrected with Fridericia's formula (QTcF) interval >480 ms
5. Chronic steroid treatment (IV or oral) or any other immunosuppressive medication (ie, prednisone >10 mg daily (QD) or the equivalent).
6. Has active other primary malignancies. Note: Participants with the following can be enrolled: Adequately resected non-melanoma skin cancer, curatively treated in situ disease, superficial cancer in the gastrointestinal tract curatively resected by endoscopic surgery, or any other solid tumors curatively treated with no evidence of recurrent disease for ≥3 years and requires no treatment.
7. Has unresolved toxicities from previous anticancer treatment, defined as toxicities (other than alopecia) not yet resolved to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0, Grade ≤1 or baseline. Note: Participants with chronic, stable Grade 2 toxicities (defined as no worsening for 1 month prior to enrollment and managed with SOC treatment) that the investigator deems related to previous anticancer treatment may be enrolled. Such toxicities may include the following:

   1. Chemotherapy-induced peripheral neuropathy
   2. Residual toxicities from prior immuno-oncology treatment:

   Grade 2 endocrinopathies (hypothyroidism, hyperthyroidism, adrenal insufficiency, hyperglycemia due to type 1 diabetes mellitus) with adequate therapy Grade 2 skin hypopigmentation (vitiligo)
8. Has known hypersensitivity to biological agents.
9. Has a history of or active autoimmune disease.

   Note: Participants with the following examples may be enrolled as an exception:
   1. Type I diabetes mellitus/hypothyroidism only requires hormone replacement.
   2. Skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment.
10. Has human immunodeficiency virus (HIV) infection. Participants must be tested for HIV viral load during the Screening Period if acceptable by local regulations or Institutional Review Boards/Independent Ethics Committees (IRBs/IECs).

    Note: For Part 2 only, the following participants will be eligible:
    1. Have CD4+ T-cell count ≥350 cells/mm3 at the time of screening.
    2. Have virologic suppression, defined as confirmed HIV RNA level below 50 or the lower limit of quantitation (below the limit of detection) at the time of screening and for at least 12 weeks before screening.
    3. Have no acquired immunodeficiency syndrome-defining opportunistic infections or conditions within the past 12 months.
    4. Are on stable antiretroviral therapy regimen, without changes in drugs or dose modification, for at least 4 weeks before trial entry (Day 1) and agree to continue antiretroviral therapy throughout the trial, as defined per institutional protocol.
11. Has active or uncontrolled hepatitis B or C infection as defined per institutional guidelines.

Note: For Part 2 only, the following participants will be eligible:

1. Hepatitis B surface antigen (HBsAg)-positive participants are eligible if they have received hepatitis B virus (HBV) antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to allocation (participants should remain on antiviral therapy throughout trial intervention and follow local guidelines for HBV antiviral therapy after completion of trial intervention).
2. Have a history of hepatitis C infection and hepatitis C virus (HCV) viral load is below the level of detection in the absence of antiviral therapy during the previous 4 weeks.
3. Have normal transaminase values, or, if liver metastases are present, abnormal transaminases with a result of AST/ALT <3 × ULN, which are not attributable to HCV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of participants with Dose-Limiting Toxicities at each dose level of DS-2243a | Up to 18 months
Part 2: Number of participants with Treatment-Emergent Adverse Events | Up to 3 years
  Descriptive statistics of treatment-emergent adverse events (TEAEs)
Part 2: Objective Response Rate | From day of first dose up to 3 years
  Objective Response Rate (ORR) as assessed by the investigator according to RECIST v1.1.

SECONDARY OUTCOMES:
Part 1: Objective Response Rate | From day of first dose up to 3 years
  ORR as assessed by the investigator according to RECIST v1.1.
Disease Control Rate | From day of first dose up to 4 years.
  Disease Control Rate (DCR) as assessed by the investigator according to RECIST v1.1.
Progression-Free Survival (PFS) | From day of first dose up to 4 years
  Progression-Free Survival (PFS) as assessed by the investigator according to RECIST v1.1.
Overall Survival | From day of first dose up to 4 years
Drug Plasma Concentration | Days 1, 2, and 3 during step-up dosing; Days 1, 2, 3, 5, 8, and 15 of Cycles 1 and 3; Day 1 of Cycle 2; and Day 1 of Cycle 4 and each subsequent cycle. A cycle may be up to 36 days.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (3):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - David H. Koch Center for Cancer Care at Memorial Sloan Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee
- UZ Leuven Europe Leuven, Leuven, Belgium
- Centre Leon Berard, Lyon, France
- Nederlands Kanker Instituut - Antoni van Leeuwenhoek Ziekenhuis (NKI-AVL), Amsterdam, Netherlands
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/